CLINICAL TRIAL: NCT02476435
Title: Depersonalization Disorder: Therapeutic Effect of Neuronavigated Repetitive Transcranial Stimulation of Right Angular Gyrus.
Brief Title: Depersonalization Disorder: Therapeutic Effect of Neuronavigated Repetitive Transcranial Stimulation
Acronym: PERSONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D14-P009
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2017-10

CONDITIONS: Depersonalization Disorder
Keywords: Depersonalization; Derealization; Embodiment; Emotional numbing; Transcranial magnetic stimulation; Angular gyrus; Temporo-parietal junction
MeSH Terms: conditions — Depersonalization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental = Active rTMS (Active Comparator): Daily rTMS with Active coil 30 minutes of 1Hz rTMS, 5 days per week, for 3 weeks
  Interventions: Device: Active rTMS
- Sham Comparator = Sham rTMS (Placebo Comparator): Daily rTMS with Sham coil 30 minutes of 1Hz rTMS, 5 days per week, for 3 weeks
  Interventions: Device: Placebo rTMS

INTERVENTIONS:
Device: Active rTMS — Strong electromagnetic fields (~2Tesla) generated briefly but repetitively (1Hz) applied for 30mins, in five sessions per week for 3 weeks
  Other Names: Strong electromagnetic fields (~2Tesla) generated briefly but repetitively (1Hz) applied for 30mins, in five sessions per week for 3 weeks
  Arms: Experimental = Active rTMS
Device: Placebo rTMS — Placebo electromagnetic fields generated briefly but repetitively applied for 30mins, in five sessions per week for 3 weeks
  Other Names: Magstim Super-Rapid2, Neuronavigation system Visor (ANT)
  Arms: Sham Comparator = Sham rTMS

SUMMARY:
The purpose of this study is to assess the therapeutic efficacy of transcranial magnetic stimulation in patients with depersonalization disorder.

DETAILED DESCRIPTION:
Depersonalization disorder is characterised by a profound disruption of self-awareness. Depersonalization symptoms may occasionally arise (30 to 70% of the population) or may become chronic in depersonalization disorder. Its prevalence is around 2.4% in the general population. This disorder is particularly resistant to pharmacological treatments. This study is a randomized, double-blind, placebo-controlled study, and the investigators are testing the therapeutic efficacy of neuronavigated repetitive Transcranial Magnetic Stimulation (TMS) of right angular gyrus in patients with depersonalization disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Outpatients aged over 18 years old
* Suffering from depersonalization disorder according to DSM IV-TR
* Patients currently on DPD medication must be at the same stable dose(s) at least 2 months and must be continued at the same dose(s) through the duration of the study.
* Patient provided informed written consent
* Patient covered by a contributory social security scheme

Controls:

* Aged over 18 years old
* Absence of a personal history of psychiatric disorders
* Provided informed written consent
* Covered by a contributory social security scheme

Exclusion Criteria:

* Patients:
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* history of neurosurgery,
* neurosurgical ventriculoperitoneal bypass valves
* personal and / or family history of seizures or epilepsy
* Dental device
* Pregnant woman
* Claustrophobic subjects
* Not cooperating or agitated patients
* Medications that reduce the seizure threshold, such as clozapine, bupropion, methadone and / or theophylline
* Alcohol abuse and / or toxic substances in the last 12 months
* Substance dependence except tobacco

Controls:

* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* neurosurgical ventriculoperitoneal bypass valves
* Claustrophobic subjects
* Pregnant woman
* Not cooperating or agitated patients
* Dental device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Cambridge Depersonalization Scale (CDS) | At 3 weeks (in the end of the treatment)
  The CDS is a comprehensive instrument containing 29 items addressing the complaints classically associated with the depersonalization syndrome. Each item is rated on two Likert scales for frequency and duration of the experience. The global score of the scale is the arithmetic sum of all items (range 0-290). High scores reflect a severe disorder.
  The improvement is defined by a 50% decrease of the scores from the Cambridge depersonalization scale
Cambridge Depersonalization Scale (CDS) | At 1 month after the treatment
  The CDS is a comprehensive instrument containing 29 items addressing the complaints classically associated with the depersonalization syndrome. Each item is rated on two Likert scales for frequency and duration of the experience. The global score of the scale is the arithmetic sum of all items (range 0-290). High scores reflect a severe disorder.
  The improvement is defined by a 50% decrease of the scores from the Cambridge depersonalization scale
Cambridge Depersonalization Scale (CDS) | At 2 months after the treatment
  The CDS is a comprehensive instrument containing 29 items addressing the complaints classically associated with the depersonalization syndrome. Each item is rated on two Likert scales for frequency and duration of the experience. The global score of the scale is the arithmetic sum of all items (range 0-290). High scores reflect a severe disorder.
  The improvement is defined by a 50% decrease of the scores from the Cambridge depersonalization scale
Cambridge Depersonalization Scale (CDS) | At 3 months after the treatment
  The CDS is a comprehensive instrument containing 29 items addressing the complaints classically associated with the depersonalization syndrome. Each item is rated on two Likert scales for frequency and duration of the experience. The global score of the scale is the arithmetic sum of all items (range 0-290). High scores reflect a severe disorder.
  The improvement is defined by a 50% decrease of the scores from the Cambridge depersonalization scale

SECONDARY OUTCOMES:
Assessment of the maintenance of therapeutic efficacy at 3 months after rTMS | At 3 months
  maintenance of reduction of at least 50% of the original score to the depersonalization scale of Cambridge.
Measurement of cerebral blood flow of the right angular gyrus and functional connectivity, measurement of cortical gyrification and anatomical connectivity | Baseline
  Anatomical MRI, ASL MRI, Resting State MRI, Diffusion MRI.
Measurement of cerebral blood flow of the right angular gyrus and functional connectivity, measurement of cortical gyrification and anatomical connectivity | Visit 3 : end of the TMS sessions (between 19 and 25 days after V2 - start of TMS)
  Anatomical MRI, ASL MRI, Resting State MRI, Diffusion MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Plaze, MD, PhD, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (2):
- France (2):
  - Saint-Antoine Hospital, Paris
  - Centre Hospitalier Sainte-Anne, Paris

REFERENCES:
- [Background] Blanke O, Ortigue S, Landis T, Seeck M. Stimulating illusory own-body perceptions. Nature. 2002 Sep 19;419(6904):269-70. doi: 10.1038/419269a. PMID 12239558
- [Background] Blanke O. Multisensory brain mechanisms of bodily self-consciousness. Nat Rev Neurosci. 2012 Jul 18;13(8):556-71. doi: 10.1038/nrn3292. PMID 22805909
- [Background] Sierra M, Berrios GE. The Cambridge Depersonalization Scale: a new instrument for the measurement of depersonalization. Psychiatry Res. 2000 Mar 6;93(2):153-64. doi: 10.1016/s0165-1781(00)00100-1. PMID 10725532
- [Background] Farrer C, Frey SH, Van Horn JD, Tunik E, Turk D, Inati S, Grafton ST. The angular gyrus computes action awareness representations. Cereb Cortex. 2008 Feb;18(2):254-61. doi: 10.1093/cercor/bhm050. Epub 2007 May 8. PMID 17490989
- [Background] Frith CD, Blakemore SJ, Wolpert DM. Abnormalities in the awareness and control of action. Philos Trans R Soc Lond B Biol Sci. 2000 Dec 29;355(1404):1771-88. doi: 10.1098/rstb.2000.0734. PMID 11205340
- [Background] Mantovani A, Simeon D, Urban N, Bulow P, Allart A, Lisanby S. Temporo-parietal junction stimulation in the treatment of depersonalization disorder. Psychiatry Res. 2011 Mar 30;186(1):138-40. doi: 10.1016/j.psychres.2010.08.022. Epub 2010 Sep 15. PMID 20837362
- [Background] Sierra M, Phillips ML, Ivin G, Krystal J, David AS. A placebo-controlled, cross-over trial of lamotrigine in depersonalization disorder. J Psychopharmacol. 2003 Mar;17(1):103-5. doi: 10.1177/0269881103017001712. PMID 12680746
- [Background] Sierra M, Baker D, Medford N, David AS. Unpacking the depersonalization syndrome: an exploratory factor analysis on the Cambridge Depersonalization Scale. Psychol Med. 2005 Oct;35(10):1523-32. doi: 10.1017/S0033291705005325. PMID 16164776
- [Background] Sierra M. Depersonalization disorder: pharmacological approaches. Expert Rev Neurother. 2008 Jan;8(1):19-26. doi: 10.1586/14737175.8.1.19. PMID 18088198
- [Background] Sierra M, David AS. Depersonalization: a selective impairment of self-awareness. Conscious Cogn. 2011 Mar;20(1):99-108. doi: 10.1016/j.concog.2010.10.018. Epub 2010 Nov 17. PMID 21087873
- [Background] Simeon D, Guralnik O, Hazlett EA, Spiegel-Cohen J, Hollander E, Buchsbaum MS. Feeling unreal: a PET study of depersonalization disorder. Am J Psychiatry. 2000 Nov;157(11):1782-8. doi: 10.1176/appi.ajp.157.11.1782. PMID 11058475
- [Background] Simeon D, Kozin DS, Segal K, Lerch B, Dujour R, Giesbrecht T. De-constructing depersonalization: further evidence for symptom clusters. Psychiatry Res. 2008 Jan 15;157(1-3):303-6. doi: 10.1016/j.psychres.2007.07.007. Epub 2007 Oct 23. PMID 17959254